CLINICAL TRIAL: NCT05206344
Title: Study on the Benefit of the Intervention of Clowns in Pediatric Oncology in the Accompaniment of Painful Acts
Brief Title: The Benefit of the Intervention of Clowns in Pediatric Oncology in the Accompaniment of Painful Acts
Acronym: ICOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Madame Valérie GAÜZES, Principal Investigator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019-A03302-55
Record Dates: First submitted 2020-10-15; First posted 2022-01-25 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without Clowns - Clowns (WC-C) (Other): Firstly a painful act without the presence of the clown duo, then in a second time the same painful act in the presence of the clown duo
  Interventions: Other: clowns
- Clowns- Without clowns (C-WC) (Other): Firstly a painful act with the presence of the clown duo, then in a seconde time, the same painful act without the presence of the clown duo
  Interventions: Other: clowns

INTERVENTIONS:
Other: clowns — presence or absence of clowns during the performance of a painful act, on pain

SUMMARY:
The diagnosis and treatment of childhood cancer involves frequent and repeated painful acts. The pediatric oncology-hematology service of Nancy's hospital innovates thanks to the involvement of clowns in the hospital. The effects of the clown's intervention corroborate the results of studies which demonstrate that when painful complaints are increased by an empathetic attitude, they are reduced by half when the child is distracted.

The main objective is to assess the impact of the presence or absence of clowns during the performance of a painful act, on pain, in children who have benefited from this act. no clowns during the performance of a painful act, on anxiety, in children who have benefited from this act.

The secondary objectives are:

* Evaluate the impact of the presence or not of clowns during the performance of a painful act, on the anxiety of the parents of the child who benefited from this act.
* Measure the perception and acceptance of the healthcare team of the presence of clowns 1 time every 3 months.
* Measure the clowns' perception of their interaction with the child, the parents and the healthcare team once every 3 months.
* Evaluate the overall impact of the clown intervention during the performance of a painful act in children on the course of the act by a "neutral" person (health manager) once every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Child virgin with experience for targeted acts during the 1st painful act or child undergoing follow-up provided that he is virgin with experience of the presence of clowns during these acts.
* Child with cancer
* Child requiring a painful act among the following 3 acts: lumbar puncture, myelogram, needle placement in an implantable chamber
* Parental authority holder (s) who have received full information on the organization of the research and who have given their written consent for the participation of their child
* Personal adhesion of the child with a view to his participation
* Presence of at least one of the two parents during act 1
* Availability of the duo of clowns for the realization of act n ° 1 if the group assigned is the group Clowns-Sans Clowns

Exclusion Criteria:

* Parents / child's refusal of clowns to intervene

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-04-08 (Estimated); Study Completion 2024-10-08 (Estimated)

PRIMARY OUTCOMES:
Change of Pain score of the patient Self Assessment Scale (VAS) | inclusion, up to 2 years
  The scale is between 0 to 100

SECONDARY OUTCOMES:
Anxiety score of the patient with modified-Yale Preoperative Anxiety Scale (m-YPAS) | inclusion, up to 2 years
  The scale is between 0 to 100 If the score is inferior to 24, the patient is considered relaxed If the score is superior to 24, the patient is considered anxious
Anxiety score of the patient with modified-Yale Preoperative Anxiety Scale (m-YPAS) | up to 8 weeks after inclusion
  The scale is between 0 to 100 If the score is inferior to 24, the patient is considered relaxed If the score is superior to 24, the patient is considered anxious
Usual Anxiety score of the parents Questionnaire State-Trait Anxiety Inventory (STAI form Y-B) | inclusion, up to 2 years
  The score is between 21 to 77 Score superior to 65 : very high anxiety Score between 56 to 65 : high anxiety Score between 46 to 55 : medium anxiety Score between 36 to 45 : low anxiety Score inferior to 35 : very low anxiety
Usual Anxiety score of the parents Questionnaire State-Trait Anxiety Inventory (STAI form Y-B) | up to 8 weeks after inclusion
  The score is between 21 to 77 Score superior to 65 : very high anxiety Score between 56 to 65 : high anxiety Score between 46 to 55 : medium anxiety Score between 36 to 45 : low anxiety Score inferior to 35 : very low anxiety
Change of Anxiety score of the parents Questionnaire State-Trait Anxiety Inventory (STAI form Y-A) | inclusion, up to 2 years
  The score is between 20 to 80 Score superior to 65 : very high anxiety Score between 56 to 65 : high anxiety Score between 46 to 55 : medium anxiety Score between 36 to 45 : low anxiety Score inferior to 35 : very low anxiety
Change of Anxiety score of the parents Questionnaire State-Trait Anxiety Inventory (STAI form Y-A) | up to 8 weeks after inclusion
  The score is between 20 to 80 Score superior to 65 : very high anxiety Score between 56 to 65 : high anxiety Score between 46 to 55 : medium anxiety Score between 36 to 45 : low anxiety Score inferior to 35 : very low anxiety
Score of perception and acceptance of the presence of clowns with the healthcare team Questionnaire | through completion of the study, an average of 2 years
  The questionnaire is composed by 19 questions The scale of each question is between 1 (not agree at all) to 4 (totally agree)
Perception score of interactions with the child, parents and the team with clowns Questionnaire | through completion of the study, an average of 2 years
  The questionnaire is composed by 12 questions The scale of each question is between 1 (not agree at all) to 4 (totally agree)
Score of evaluation of the overall impact of the presence or not of a clown Questionnaire | through completion of the study, an average of 2 years
  The observation gris is composed by 14 questions

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Chastagner, Study Director — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Nancy, France